CLINICAL TRIAL: NCT06671756
Title: The Metabolic Response to Fructose Ingestion
Brief Title: Metabolic Effects of Fructose Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Mark Andrew Herman, Associate Professor; Chief, Section of Endocrinology, Diabetes, and Metabolism, Medicine, Baylor College of Medicine, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: H55353
Record Dates: First submitted 2024-10-24; First posted 2024-11-04 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Healthy
Keywords: Fructose; Metabolism; Soluble Leptin Receptor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fructose First, Glucose Second (10 participants) (Experimental): Participants will first consume 75g of fructose in 225ml of water. Blood samples will be taken at specific intervals to measure metabolic responses. After 2 weeks, they will consume 75g of glucose in 225ml of water, with blood samples taken at the same intervals.
  Interventions: Dietary Supplement: Fructose Ingestion; Dietary Supplement: Glucose Ingestion
- Glucose First, Fructose Second (10 participants) (Experimental): Participants will first consume 75g of glucose in 225ml of water, followed by the same blood sampling schedule. After 2 weeks, they will switch to 75g of fructose, with blood samples taken at the same intervals.
  Interventions: Dietary Supplement: Fructose Ingestion; Dietary Supplement: Glucose Ingestion

INTERVENTIONS:
Dietary Supplement: Fructose Ingestion — Participants will consume a beverage containing 75g of fructose dissolved in 225ml of water.
Dietary Supplement: Glucose Ingestion — Participants will consume a beverage containing 75g of glucose dissolved in 225ml of water.

SUMMARY:
The goal of this clinical trial is to learn how fructose ingestion affects metabolic factors in healthy adults aged 18-64, with a BMI between 19 and 30 kg/m², of any sex or gender. Specifically, the study aims to examine the impact of fructose compared to glucose on circulating metabolic factors including the soluble leptin receptor.

The main questions it aims to answer are:

How does fructose ingestion influence levels of circulating metabolic markers, including the soluble leptin receptor? Does fructose consumption have different metabolic effects compared to glucose?

Participants will:

Complete a screening phone call to review their health history and eligibility.

Attend two in-person visits at least two weeks apart, where they will:

Fast for 8 hours beforehand. Consume a beverage containing either 75g of fructose or glucose. Have blood drawn at regular intervals for up to 5 hours after consumption to measure circulating levels of metabolic markers.

ELIGIBILITY:
Inclusion Criteria:

* Age: Participants must be between 18 and 64 years old.
* BMI: Participants must have a Body Mass Index (BMI) between 19 and 30 kg/m² (healthy weight to slightly overweight).
* Health Status: Participants must be healthy volunteers with no significant medical conditions.
* Sex/Gender: Both males and females are eligible to participate.

Exclusion Criteria:

* Known significant medical illness, any medications except oral contraceptives, history of fructose intolerance, pregnancy. We will not enroll BCM Medical students or individuals who work directly for any of the study investigators.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in Circulating Levels of Soluble Leptin Receptor After Fructose Ingestion | From baseline (Day 0) to 300 minutes post-ingestion.
  The study will measure changes in the blood levels of soluble leptin receptor (ng/mL) following fructose ingestion. These levels will be assessed at multiple time points-baseline (0 minutes), 30 minutes, 60 minutes, 120 minutes, 180 minutes, 240 minutes, and 300 minutes post-ingestion-to evaluate how fructose affects their concentrations compared to baseline levels and glucose ingestion.

SECONDARY OUTCOMES:
Change in Circulating Levels of fibroblast growth factor 21(FGF 21) | From baseline (0 minutes) to 300 minutes post-ingestion.
  The study will assess changes in FGF21 levels (pg/mL) in response to fructose and glucose ingestion. FGF21 levels will be measured at specific time points-baseline (0 minutes), 30 minutes, 60 minutes, 120 minutes, 180 minutes, 240 minutes, and 300 minutes post-ingestion-to explore the effects of these sugars.
Change in Circulating Insulin Levels | From baseline (0 minutes) to 300 minutes post-ingestion.
  The study will evaluate changes in insulin levels (µIU/mL) following fructose and glucose ingestion. Insulin levels will be measured at baseline (0 minutes), 30 minutes, 60 minutes, 120 minutes, 180 minutes, 240 minutes, and 300 minutes post-ingestion to assess how these sugars affect insulin secretion and metabolic regulation.
Change in Triglyceride Levels | From baseline (0 minutes) to 300 minutes post-ingestion.
  The study will measure changes in circulating triglyceride levels (mg/dL) to explore how fructose and glucose ingestion affect lipid metabolism. Triglyceride levels will be measured at baseline (0 minutes), 30 minutes, 60 minutes, 120 minutes, 180 minutes, 240 minutes, and 300 minutes post-ingestion.
Change in Cholesterol Levels | From baseline (0 minutes) to 300 minutes post-ingestion.
  The study will assess changes in total cholesterol levels ((mg/dL) following fructose and glucose ingestion to evaluate potential effects on cholesterol metabolism. Cholesterol levels will be measured at baseline (0 minutes), 30 minutes, 60 minutes, 120 minutes, 180 minutes, 240 minutes, and 300 minutes post-ingestion.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor St. Luke's Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data will be shared with academic investigators upon request.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: This information will be available for 5 years following publication of the study.
Access Criteria: Academic investigators upon request to the study's PI.

REFERENCES:
- [Background] Fisher FM, Kim M, Doridot L, Cunniff JC, Parker TS, Levine DM, Hellerstein MK, Hudgins LC, Maratos-Flier E, Herman MA. A critical role for ChREBP-mediated FGF21 secretion in hepatic fructose metabolism. Mol Metab. 2016 Nov 23;6(1):14-21. doi: 10.1016/j.molmet.2016.11.008. eCollection 2017 Jan. PMID 28123933
- [Background] Katz LS, Baumel-Alterzon S, Scott DK, Herman MA. Adaptive and maladaptive roles for ChREBP in the liver and pancreatic islets. J Biol Chem. 2021 Jan-Jun;296:100623. doi: 10.1016/j.jbc.2021.100623. Epub 2021 Apr 2. PMID 33812993
- [Background] Kim MS, Krawczyk SA, Doridot L, Fowler AJ, Wang JX, Trauger SA, Noh HL, Kang HJ, Meissen JK, Blatnik M, Kim JK, Lai M, Herman MA. ChREBP regulates fructose-induced glucose production independently of insulin signaling. J Clin Invest. 2016 Nov 1;126(11):4372-4386. doi: 10.1172/JCI81993. Epub 2016 Sep 26. PMID 27669460
- [Background] Sargsyan A, Doridot L, Hannou SA, Tong W, Srinivasan H, Ivison R, Monn R, Kou HH, Haldeman JM, Arlotto M, White PJ, Grimsrud PA, Astapova I, Tsai LT, Herman MA. HGFAC is a ChREBP-regulated hepatokine that enhances glucose and lipid homeostasis. JCI Insight. 2023 Jan 10;8(1):e153740. doi: 10.1172/jci.insight.153740. PMID 36413406
- [Background] Herman MA, Birnbaum MJ. Molecular aspects of fructose metabolism and metabolic disease. Cell Metab. 2021 Dec 7;33(12):2329-2354. doi: 10.1016/j.cmet.2021.09.010. Epub 2021 Oct 6. PMID 34619074